CLINICAL TRIAL: NCT00996827
Title: Ultraviolet Light Exposure and Immunosuppression in Cutaneous Melanoma
Status: Terminated | Type: Observational
Why Stopped: Sufficient samples collected when 73% of target enrollment was reached.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0815
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Melanoma
Keywords: Melanoma; Skin cancer; Vitamin D; Vitamin D receptor; Sunlight; Cytokine
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serum samples will be collected to evaluate the immune status of these patients.
  * Serum cytokine profiles
  * Whole blood samples - lymphocyte sub-populations from fresh, refrigerated whole blood samples. Whole blood samples will be used to extract DNA and RNA material. The remaining DNA for future research related to cytokine gene and vitamin D receptor single nucleotide polymorphisms studies of the Molecular Epidemiology Laboratory
  * H & E slides will be evaluated by our collaborating pathologist to validate diagnoses and Breslow thickness
  * Formalin-fixed paraffin embedded blocks will be sectioned and stained for immunohistochemistry
  * One slide will be prepared from the skin block to evaluate the presence of solar elastosis in relation to UV exposure
Oversight: Data Monitoring Committee: No

SUMMARY:
This project seeks to understand differences in the serum vitamin D levels and immune status in cutaneous malignant melanoma patients with different UV exposure histories in New Mexico.

DETAILED DESCRIPTION:
It is well established that ultraviolet radiation (UV) exposure is related to the development of melanoma. There is also evidence that immune reactions are altered after UV exposure in the skin (locally) and perhaps throughout the body (systemically). Additionally, while the role of vitamin D and melanoma development has not been fully established, UV-B exposure is essential for vitamin D production in the skin. Increased sun exposure is also related to the presence of solar elastosis, which might protect (1) or improve survival from melanoma. Thus, melanoma represents a unique model for studying UV exposure, the immune system, and vitamin D. Malignant melanoma is an antigenic cancer; therefore, the role of UV exposure-induced immunosuppression and vitamin D production in the recognition, destruction and growth inhibition of cancerous melanocytes is worth further study.

To underscore the importance of this project, the Scientific Advisory Committee of the Melanoma Research Foundation and the Steering Committee of the Society of Melanoma Research have indicated a need to collect more human data on the host immune response mechanisms in melanoma and also to focus on the skin as a whole microenvironment, moving away from only in vitro experiments.

ELIGIBILITY:
Inclusion Criteria:

* Resident of New Mexico
* Age between the 1 and 95
* Newly diagnosed with cutaneous invasive melanoma; any stage permitted (ICDO C44.0-9) between September 1, 2008 and December 31, 2011.
* SSM (superficial spreading melanoma) and NM (nodular melanoma) histological subtypes are allowed
* Access to a telephone or be able to participate in a personal interview at the clinic
* Physically and mentally competent to complete a 1-hour telephone or personal interview

Exclusion Criteria:

* Ocular melanoma, LMM (lentigo maligna melanoma) or ALM (acral lentigo melanoma), and mucosal melanoma cases.
* No access to a telephone or is not able to meet with the interviewer.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have recieved interferon or IL-2 therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
• Evaluate serum 25(OH)-vitamin D concentrations. • Detect the presence of solar elastosis and local immunosuppression in skin biopsy samples • Assess the role of the systemic humoral immune response | 1 year

SECONDARY OUTCOMES:
• Evaluate cellular immunological changes of peripheral lymphocyte subpopulations • Sequence chromosome 6 from blood DNA samples of the patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Montasur Shaheen, MD, Principal Investigator — University of New Mexico; Marianne Berwick, PhD, Study Chair — University of New Mexico Cancer Center
Locations (2):
- United States (2):
  - Lovelace Women's Hospial, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org